CLINICAL TRIAL: NCT06419751
Title: Research on the Effect of Lifestyle Intervention Combined With Wearable Devices Based on Different Exercise on Vascular Health
Brief Title: the Effects of Different Exercise on Vascular Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-ZX067
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Mind-body Exercise; Vascular Health; M-health; Cardiac Rehabilitation
Keywords: m-health; mind-body exercise; cardiac rehabilitation; arterial stiffness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Study participants were given training on dietary patterns, regular monitoring and follow-up through apps and wearable devices, and no forced exercise measures were performed.
- Combined Exercise Group (Active Comparator): Study participants were given training on dietary patterns, regular monitoring and follow-up through apps and wearable devices.Based on the status of the study participants and the results of the cardiopulmonary exercise test, the investigators prescribe moderate-intensity aerobic exercise combined with resistance exercise
  Interventions: Behavioral: Regular exercise
- Mind-body Exercise Group (Experimental): Study participants were given training on dietary patterns, regular monitoring and follow-up through apps and wearable devices.A standardized Baduanjin exercise program consists of eight postures, each training time is about 30 minutes (including 10 min warm-up, 2 times of Baduanjin, and 10 min of relaxation), 5 days/week, a total of 12 weeks.
  Interventions: Behavioral: Baduanjin

INTERVENTIONS:
Behavioral: Regular exercise — Based on the study participant's status and exercise assessment, the investigators prescribe moderate-intensity aerobic exercise combined with resistance exercise. Before each exercise, preparatory activities (10min), 20-30min moderate-intensity aerobic exercise, finishing activities (10min) at the end, 5 days/week, for 12 weeks, and at the same time, choose non-consecutive 3 days of resistance training in 5 aerobic training sessions to increase resistance training (choose 1~2 muscle groups each time, 4~5 movements, repeat each action 8~12 times, repeat 2~3 sets)
  Arms: Combined Exercise Group
Behavioral: Baduanjin — A professional therapist instructed the participants to learn and train Baduanjin before the intervention, and a standardized Baduanjin exercise program included eight postures, each training time was about 50 minutes (including 10 min of warm-up, 2 times of Baduanjin, and 10 min of relaxation), 5 days/week, a total of 12 weeks
  Arms: Mind-body Exercise Group

SUMMARY:
To explore the effect of smart app and wearable-based lifestyle intervention management on vascular health, comparing different exercise with the improvement of vascular arterial stiffness. The accuracy and consistency evaluation of smart wearable devices in screening for vascular health risks were also discussed.

DETAILED DESCRIPTION:
This study intends to carry out a randomized controlled trial to dynamically monitor a variety of cardiovascular parameters in people with high risk of vascular health, using wearable devices and artificial intelligence-assisted health management platform, and provide intelligent lifestyle intervention programs with different exercise.By observing the improvement of vascular health in the study population, the management effect of intelligent lifestyle intervention on high-risk groups of vascular health was evaluated. It is expected that through comprehensive lifestyle intervention based on smart wearable devices, early prevention and control of arteriosclerosis can be achieved, the level of hospital health management will be improved, and more physical health and health economic benefits will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and < 60 years old;
2. cfPWV>10m/s;
3. Those who have 1 intelligent communication device and can use it proficiently (Android mobile phone is preferred);
4. People who have lived and/or worked relatively steadily in the past 6 months;
5. Signed informed consent.

Exclusion Criteria:

1. Moderate to severe obesity (≥30kg/m^2);
2. Acute myocardial infarction, acute tachyarrhythmia, pulmonary edema, severe aortic stenosis and other serious circulatory respiratory diseases and acute cardiovascular and cerebrovascular diseases;
3. severe essential hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg) or poorly controlled essential hypertension;
4. Patients with secondary hypertension, acute hypertension, subacute hypertension and hypertensive encephalopathy;
5. Significant arrhythmia (atrial fibrillation, etc.);
6. Patients with atherosclerotic cardiovascular diseases, such as coronary heart disease, severe peripheral atherosclerotic diseases, etc.;
7. Type 1 diabetes, uncontrolled type 2 diabetes or other diseases affecting carbohydrate metabolism;
8. Severe stenosis of the carotid and/or femoral arteries (resulting in significant abnormalities in the blood flow spectrum); Those who have anatomical abnormalities of the aorta and major branches and cannot complete PWV detection;
9. Cancer and other major comorbidities affecting arterial blood pressure;
10. Those who are unable to exercise due to fractures, joint instability and other physical diseases or diseases affecting the locomotor system;
11. Those who have involuntary physical movements due to mental illness, epilepsy or other diseases;
12. Those who have a pacemaker installed;
13. Pregnant/trying to conceive;
14. Patients with allergies, limb trauma or skin diseases who cannot cooperate with the completion of ABI and baPWV index examinations;
15. Those who have undergone or plan to have bariatric surgery in the next 12 months;
16. Those who have participated in other clinical studies in the past 3 months;
17. Refusal to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cervical femoral pulse wave velocity（cfPWV） | baseline,3months,6months,9 months
  The cardio-cerebrovascular and aortic function detector (Campura, France, model: Complior Analyse) was used to measure cfPWV, and the study participants were in a supine position, lying flat on the pillow, with their palms up on their sides of the body, so that their whole body was relaxed and rested for about 3 minutes. PWV can reflect arterial stiffness, and the European Society of Cardiology recommends cfPWV >10 m/s as the definitive threshold for assessing arterial functional changes in hypertension.We monitored cfPWV at baseline,3,6,9 months of the study.

SECONDARY OUTCOMES:
Brachi-ankle pulse wave velocity（baPWV） | baseline,3months,6months,9 months
  The blood pressure of the limbs is measured with the Omron arteriosclerosis detector, and the pulse conduction velocity (baPWV) and ankle-brachial index (ABI) are calculated to automatically evaluate the degree of arteriosclerosis and blood vessel blockage. Positive criteria for baPWV: ≥1400 cm/s or baPWV% ≥ 19% is arteriosclerosis. Lower extremity vascular occlusion (ABI positive criteria): ≤0.9 for peripheral arterial stenosis and ≤0.5 for possible peripheral arterial occlusion.We monitored baPWV at baseline,3,6,9 months of the study.
blood pressure | baseline,3months,6months,9 months
  Blood pressure indicator: systolic blood pressure and diastolic blood pressure.We monitored blood pressure at baseline,3,6,9 months of the study.
body weight | baseline,3months,6months,9 months
  Using bioelectrical impedance analysis to monitor body weight,weight and height will be combined to report BMI in kg/m^2.We monitored body composition at baseline,3,6,9 months of the study.
Lipid metabolism parameters: TC(mmol/L), TG(mmol/L), HDL-C(mmol/L), LDL-C(mmol/L) | baseline,3months,6months,9 months
  Lipid metabolism indicators: total cholesterol , triglyceride , high density lipoprotein cholesterol, low density lipoprotein cholesterol.We monitored lipid metabolism parameters at baseline,3,6,9 months of the study.
Physical fitness | baseline,3months,6months,9 months
  The measurement of muscle strength, balance and flexibility is completed by the rehabilitation therapist, mainly including: (1) upper limb muscle strength test (dumbbell arm curl test); (2) Lower limb muscle strength test (chair standing and sitting test); (3) balance ability test; (4) Lower limb flexibility assessment (chair sitting body forward bending test); (5) Upper limb flexibility assessment (two-hand dorsum extension test). Participants were observed for changes at baseline, 3,6,9 months.
Vascular Health Index | baseline,3months,6months,9 months
  The PWV was analyzed by the smart watch through ECG (electrocardiogram) and PPG (photoplethysmography) sensors to evaluate the degree of vascular elasticity, and the vascular health index and evaluation were obtained, and the results were divided into low-risk, medium-risk, and high-risk.
Application adherence | baseline,3months,6months,9 months
  Study participants who received remote lifestyle interventions through the app, completed all exercise training content per week, or clocked in ≥ exercise 3 times were considered to have good compliance; Those who check in < exercise 3 times a week are considered to have poor compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Feng, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital